CLINICAL TRIAL: NCT07290569
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Dose-range Finding Study of ORKA-001 in Participants With Moderate-to-Severe Plaque Psoriasis
Brief Title: Dose Ranging Study of ORKA-001 in Patients With Moderate-to-Severe Plaque Psoriasis
Acronym: EVERLAST-B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oruka Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORKA-001-114
Record Dates: First submitted 2025-12-16; First posted 2025-12-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis
Keywords: Phase 2; ORKA-001; Plaque psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- (Induction Period - Arm 1) ORKA-001 (Experimental): Participants will receive 37.5 mg ORKA-001 per protocol Induction regimen.
  Interventions: Drug: ORKA-001
- (Induction Period - Arm 2) ORKA-001 (Experimental): Participants will receive 300 mg ORKA-001 per protocol Induction regimen.
  Interventions: Drug: ORKA-001
- (Induction Period - Arm 3) ORKA-001 (Experimental): Participants will receive 600 mg ORKA-001 per protocol Induction regimen.
  Interventions: Drug: ORKA-001
- (Induction Period - Arm 4) Placebo (Placebo Comparator): Participants will receive Placebo per protocol Induction regimen.
  Interventions: Other: Placebo
- (Maintenance Period - Arm 1) ORKA-001 (Experimental): Participants will receive 300 mg ORKA-001 per protocol Maintenance regimen, based on protocol defined response.
  Interventions: Drug: ORKA-001
- (Maintenance Period - Arm 2) ORKA-001 (Experimental): Participants will receive 600 mg ORKA-001 per protocol Maintenance regimen, based on protocol defined response.
  Interventions: Drug: ORKA-001
- (Maintenance Period - Arm 3) Placebo (Placebo Comparator): Participants will receive Placebo per protocol Maintenance regimen, based on protocol defined response.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ORKA-001 — ORKA-001 administered by subcutaneous (SC) injection
  Arms: (Induction Period - Arm 1) ORKA-001; (Induction Period - Arm 2) ORKA-001; (Induction Period - Arm 3) ORKA-001; (Maintenance Period - Arm 1) ORKA-001; (Maintenance Period - Arm 2) ORKA-001
Other: Placebo — Placebo administered by subcutaneous (SC) injection
  Arms: (Induction Period - Arm 4) Placebo; (Maintenance Period - Arm 3) Placebo

SUMMARY:
This is a multicenter, randomized, double-blinded, placebo-controlled, dose-range finding study to evaluate the efficacy and safety of ORKA-001 in adult participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, placebo-controlled, dose ranging study designed to identify the optimal induction dosing regimen of ORKA-001 in approximately 160 adult participants with moderate-to-severe plaque psoriasis.

The study will evaluate the efficacy and safety of 3 induction dosing regimens of ORKA-001 compared to placebo and will include 3 maintenance regimens.

The study will consist of 4 periods:

* Screening Period of up to 6 weeks
* Induction Period of up to 28 weeks (Day 1 [Baseline] to Week 28)
* Maintenance Period of up to approximately 72 weeks (Week 28 to Week 100)
* Post-treatment Follow-up Period: Participants will have the option to enter the open-label extension (OLE) study. Participants who opt out of the OLE study and/or withdraw from the study must be followed for 48 weeks after the End of Treatment (EOT)/Early Termination (ET) visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥ 18 years of age
2. Have a diagnosis of plaque psoriasis for > 6 months
3. Have moderate-to-severe chronic plaque psoriasis defined as:

   1. BSA ≥ 10%, and
   2. PASI ≥ 12, and
   3. IGA score of ≥ 3 on a 5-point scale
4. Candidate for systemic therapy or phototherapy
5. Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

1. Nonplaque forms of psoriasis (including guttate, erythrodermic, or pustular) or drug-induced psoriasis
2. Significant history or clinical manifestation of any metabolic, other dermatological, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, respiratory, endocrine, or psychiatric disorder, or any infectious disease
3. History of malignancy, except for non-melanoma skin cancer or cancer curatively treated ≥ 5 years, without evidence of recurrence
4. A known hypersensitivity to any components of the ORKA-001 drug product
5. Women who are breastfeeding or plan to breastfeed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving 100% Reduction in PASI Score at Week 16 | Week 16
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).

SECONDARY OUTCOMES:
Proportion of Participants Who Achieve an IGA = 0 (Clear) at Week 16 | Week 16
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Achieving 90% Reduction in PASI Score at Week 16 | Week 16
  Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Proportion of Participants Who Achieve an IGA = 0 (Clear) or 1 (Almost Clear) at Week 16 | Week 16
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Maintaining 100% Reduction in PASI Score at Week 100 | Week 100
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Proportion of Participants Maintaining an IGA = 0 (Clear) at Week 100 | Week 100
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Maintaining 90% Reduction in PASI Score at Week 100 | Week 100
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Proportion of Participants Maintaining an IGA = 0 (Clear) or 1 (Almost Clear) at Week 100 | Week 100
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Maintaining 75% Reduction in PASI Score at Week 100 | Week 100
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Incidence of Treatment-emergent Adverse Events (TEAEs) and TEAEs of Special Interest (TEAESIs) | Day 1 through Week 100
  Incidence of treatment adverse events, treatment adverse events of special interest, and clinically significant changes from baseline in vital signs, clinical laboratory parameters and electrocardiograms

CONTACTS AND LOCATIONS:
Locations (19):
- United States (13):
  - Oruka Therapeutics Investigative Site, Phoenix, Arizona
  - Oruka Therapeutics Investigative Site, North Little Rock, Arkansas
  - Oruka Therapeutics Investigative Site, Los Angeles, California
  - Oruka Therapeutics Investigative Site, Coral Gables, Florida
  - Oruka Therapeutics Investigative Site, Rolling Meadows, Illinois
  - Oruka Therapeutics Investigative Site, Plainfield, Indiana
  - Oruka Therapeutics Investigative Site, Kew Gardens, New York
  - Oruka Therapeutics Investigative Site, Mason, Ohio
  - Oruka Therapeutics Investigative Site, Portland, Oregon
  - Oruka Therapeutics Investigative Site, Frisco, Texas
  - Oruka Therapeutics Investigative Site, Houston, Texas
  - Oruka Therapeutics Investigative Site, Webster, Texas
  - Oruka Therapeutics Investigative Site, Norfolk, Virginia
- Canada (6):
  - Oruka Therapeutics Investigative Site, Surrey, British Columbia
  - Oruka Therapeutics Investigative Site, Fredericton, New Brunswick
  - Oruka Therapeutics Investigative Site, Ajax, Ontario
  - Oruka Therapeutics Investigative Site, Peterborough, Ontario
  - Oruka Therapeutics Investigative Site, Montreal, Quebec
  - Oruka Therapeutics Investigative Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided